CLINICAL TRIAL: NCT02992808
Title: Follicular Fluid, Serum Endocrine Profile Following Stimulation With Recombinant Gonadotropins or Highly Purified Human Menopausal Gonadotropin During GnRH-antagonist Protocol
Brief Title: Androgenic Profile Following Controlled Ovarian Stimulation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Eran Zilberberg, Senior physician, Infertility & IVF Unit, Department of Obstetrics & Gynecology, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-16-3516-EZ-CTIL
Record Dates: First submitted 2016-12-11; First posted 2016-12-14 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Infertility, Female
Keywords: IVF; Ovarian stimulation; Androgenic profile; Follicular fluid; Recombinant gonadotropins; human menopausal gonadotropin
MeSH Terms: conditions — Infertility, Female | interventions — pergoveris; Luteinizing Hormone, beta Subunit; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recombinant preparations (Active Comparator)
  Interventions: Drug: recombinant gonadotropins
- HP-HMG (Active Comparator): Highly purified human menopausal gonadotropin
  Interventions: Drug: HP-HMG

INTERVENTIONS:
Drug: recombinant gonadotropins
  Other Names: Pergoveris & Luveris
  Arms: Recombinant preparations
Drug: HP-HMG
  Other Names: Menopur
  Arms: HP-HMG

SUMMARY:
In this study the investigators will try to discover whether there is a difference for any of the stimulation preparations - recombinant FSH + recombinant LH (pergoveris & luveris) vs. human menopausal gonadotropin (menopur) during GnRH-antagonist cycles in the meaning of androgenic hormones profile. The study question is whether using recombinant LH will result in different follicular hormonal milieu, serum endocrine profile or IVF outcomes than using highly purified urinary gonadotropins with hCG mimicking LH activity.

DETAILED DESCRIPTION:
ABSTRACT:

The optimal controlled ovarian stimulation (COH) protocol is yet to be decided and most probably there is no right protocol that is optimal for all patients.

The role of luteinizing hormone (LH) administration during controlled ovarian stimulation (COH) is widely debated in the current medical literature.

Until recently the only source for exogenous LH activity was HMG preparations, however, in the past few years an advancement in the field of recombinant technology resulted in recombinant preparations of LH. In contrast to LH activity in HMG which is mainly due to hCG rather than from LH, using r-LH provides true, consistent and precise LH activity.

In the past years few papers were published about the difference between recombinant follicle stimulating hormone (r-FSH) and menotropins but there is still a need for researching the different effects of gonadotropins preparations and in particular the effect of LH administration during COH in the manner of follicular endocrine characteristics, embryo quality and pregnancy outcomes.

In the present study the investigators aim to elucidate whether there is a difference for any of the stimulation preparations - recombinant FSH + recombinant LH (pergoveris & luveris) vs. human menopausal gonadotropin (menopur) during GnRH-antagonist cycles. The study question is whether using recombinant LH will result in different follicular hormonal milieu, serum endocrine profile or IVF outcomes than using highly purified urinary gonadotropins with hCG mimicking LH activity.

In the relevant medical literature there is one prospective study dealing with the same question, but, during long-GnRH-agonist cycles. In the aforementioned paper there were no significant differences between the two stimulation preparations.

MATERIALS & METHODS:

Study design - A non-intervention observational trial. Primary endpoint - Serum & follicular fluid hormonal profile during COH (FSH, LH, progesterone, estradiol, testosterone, androstendione, 17-OH progesterone) Secondary endpoints - Implantation rate, clinical pregnancy, # of follicles, # of oocytes, # of embryos, top quality embryos.

Study sample - 100 patients undergoing COH for IVF using the GnRH-antagonist protocol Inclusion criteria - 20-40 years old IVF patients, BMI 19-35 undergoing their 1-4 IVF cycle.

Exclusion criteria - Suspected PCOS, history of OHSS, Patients who had a chronic illness or were receiving chronic medical treatment will be excluded.

Gonadotropin preparations -

1. As HP-HMG we will use Menopur© (menotropins for injection, FERRING) which contains equal amount of FSH & LH.
2. As the recombinant preparation we will use Pergoveris© (follitropin alfa/lutropin alfa, MERCK SERONO) which contains 150 units of FSH + 75 units of LH and Luveris© (lutropin alfa, MERCK SERONO) which is LH only preparation.

The patients - The study population will consist of all consecutive eligible patients attending the IVF unit of our department for treatment of infertility. The study required no modification of our routine, flexible, multi-dose GnRH antagonist protocol.

Briefly, after the presence of quiescent ovaries on transvaginal ultrasound and low serum E2 level were confirmed on day 2/3 of menstruation, recombinant FSH - Gonal-F© (follitropin alfa; MERCK SERONO) will be administered subcutaneously at a starting dose of 150-300 IU, depending on patient's age and/or ovarian responsiveness in previous cycles. The gonadotropin dosage will be adjusted individually according to serum E2 levels and vaginal ultrasound measurements of follicular diameter, obtained every one or two days. LH will be added to the protocol as urinary preparation Menopur© (menotropins for injection, FERRING) or as recombinant preparations - Pergoveris© (follitropin alfa/lutropin alfa, MERCK SERONO) with or without Luveris© (lutropin alfa, MERCK SERONO). GnRH-antagonist - Cetrotide© (cetrorelix, MERCK SERONO), 0.25 mg daily subcutaneously, will be added when the leading follicle reached 14-16 mm diameter, and will be continued until the day of ovulation triggering. When at least three mature (>17 mm) follicles will be obtained, patients will receive an injection of either Ovitrelle© 250 mcg (Choriogonadotropin alfa, MERCK SERONO) or GnRH-agonist - Decapeptyl© 0.2 mg (Triptorelin acetate, FERRING).

In summary, for the purpose of the study, in addition to the routine monitoring during the COH cycle, blood samples will be drawn to determine the hormonal profile (E2, progesterone), levels of serum androgens, namely, testosterone, androstendione, 17-OH progesterone and LH and FSH: (1) day 1-3 of menstruation (Day-S); (2) day of or prior to hCG administration (Day-hCG); and (3) day of ovum pick-up (Day-OPU).

Moreover, pooled follicular fluid will be collected after oocytes retrieval (fluid destined to be discarded) and will be examined for hormonal profile (FSH, LH, progesterone, estradiol, testosterone, androstendione, 17-OH progesterone).

To note - participation in this study WILL NOT change the COH treatment.

Statistics - The chi-squared test and analysis of variance (ANOVA) will be applied to detect statistically significant differences among the groups with regard to proportions or means. A two-sided P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women between 20-40 years of age
* BMI 19-35
* undergoing their 1-4 IVF cycle

Exclusion Criteria:

* Suspected PCOS
* History of OHSS
* Patients who had a chronic illness or were receiving chronic medical treatment

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Serum hormonal profile | (1) day 1-3 of menstruation (Day-S); (2) day of or prior to hCG administration (Day-hCG); and (3) day of ovum pick-up (Day-OPU).
  Hormonal profile = FSH, LH, progesterone, estradiol, testosterone, androstendione, 17-OH progesterone
Follicular fluid hormonal profile | Ovum pick up day
  Hormonal profile = FSH, LH, progesterone, estradiol, testosterone, androstendione, 17-OH progesterone

SECONDARY OUTCOMES:
Implantation rate | About three weeks after embryo transfer
  Number of gestational sacs on US exam / number of retrieved embryos
Clinical pregnancy | About three weeks after embryo transfer
  Number of cases with gestational sac per US exam / cases of embryo transfer
Biochemical pregnancy | About two weeks after embryo tranfer
  Positive BHCG test
Ongoing pregnancy | 10-12 weeks after embryo tranfer
  Number of viable pregnancies at about 10-12 weeks of gestation
Live birth rate | Until about 40 weeks after embryo transfer
  Number of pregnancies ended in a live birth
Number of follicles | During stimulation - one-two dayes before ovum pick-up
  Larger than 14 mm follicles per US
Number of oocytes retrieved | 1 day right after ovarian pick-up
  Number of oocytes retrieved during ovarian pick-up
Number of embryos | About 3 days after OPU (ovum pick-up)
  Number of developing embryos in the laboratory
Number of top quality embryos | 3 days after OPU
  The number of day 3 embryos with 7-8 cells with less than 15% fragmentation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen AN, Devroey P, Arce JC. Clinical outcome following stimulation with highly purified hMG or recombinant FSH in patients undergoing IVF: a randomized assessor-blind controlled trial. Hum Reprod. 2006 Dec;21(12):3217-27. doi: 10.1093/humrep/del284. Epub 2006 Jul 27. PMID 16873892
- [Background] Devroey P, Pellicer A, Nyboe Andersen A, Arce JC; Menopur in GnRH Antagonist Cycles with Single Embryo Transfer Trial Group. A randomized assessor-blind trial comparing highly purified hMG and recombinant FSH in a GnRH antagonist cycle with compulsory single-blastocyst transfer. Fertil Steril. 2012 Mar;97(3):561-71. doi: 10.1016/j.fertnstert.2011.12.016. Epub 2012 Jan 13. PMID 22244781
- [Background] Van Wely M, Westergaard LG, Bossuyt PM, Van der Veen F. Human menopausal gonadotropin versus recombinant follicle stimulation hormone for ovarian stimulation in assisted reproductive cycles. Cochrane Database Syst Rev. 2003;(1):CD003973. doi: 10.1002/14651858.CD003973. PMID 12535497
- [Background] Requena A, Cruz M, Ruiz FJ, Garcia-Velasco JA. Endocrine profile following stimulation with recombinant follicle stimulating hormone and luteinizing hormone versus highly purified human menopausal gonadotropin. Reprod Biol Endocrinol. 2014 Jan 29;12:10. doi: 10.1186/1477-7827-12-10. PMID 24476504
- [Background] Revelli A, Pettinau G, Basso G, Carosso A, Ferrero A, Dallan C, Canosa S, Gennarelli G, Guidetti D, Filippini C, Benedetto C. Controlled Ovarian Stimulation with recombinant-FSH plus recombinant-LH vs. human Menopausal Gonadotropin based on the number of retrieved oocytes: results from a routine clinical practice in a real-life population. Reprod Biol Endocrinol. 2015 Jul 25;13:77. doi: 10.1186/s12958-015-0080-6. PMID 26209525